CLINICAL TRIAL: NCT01262144
Title: A Study to Evaluate the Value of SUV-Max in PET-FDG in Predicting Outcome of Surgery Vis a Vis Need for Radiotherapy
Brief Title: SUV Max as Predictor of Outcome in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Amit Amnon, director, gynecologic oncology unit, Rambam Health Care Campus
Other Study IDs: 421CTIL
Record Dates: First submitted 2010-11-23; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; PET CT; SUV Max
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case group
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy for cervical cancer

SUMMARY:
Cervical Cancer is staged clinically, not surgically. Patients in whom an extensive disease is identified are not usually eligible for surgery. PET-CT is used to support staging. However, some patients received surgery after staging and subsequently require radio/chemotherapy due to findings on operation.

This study will attempt to find a correlation between SUV-Max on PET-CT and subsequent outcomes i.e. need for adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* having stating PET-CT stored on site
* treated with surgery

Exclusion Criteria:

* not eligible for surgery based on PET-CT, clinical stage

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females age 18-80, diagnosed with cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-08

PRIMARY OUTCOMES:
Administration of adjuvant therapy | immediately following surgery

SECONDARY OUTCOMES:
Overall survival | surgery - present day

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Amit, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, City, Haifa District, Israel